CLINICAL TRIAL: NCT04107220
Title: Comparison of BNP and NT-proBNP in the Management of Patients With Chronic and Acute Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Alere, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN0014
Record Dates: First submitted 2016-08-30; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Heart Failure
Keywords: BNP; NT-proBNP; ARNI; Sacubitril/Valsartan
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one arm (Other): One arm study patients where NT-proBNP and BNP tests will be monitored.
  Interventions: Drug: Sacubitril/Valsartan

INTERVENTIONS:
Drug: Sacubitril/Valsartan — Effect of Sacubitril/Valsartan on BNP and NT-proBNP
  Other Names: Entresto

SUMMARY:
The purpose of this study is to compare the changes in B-type Natriuretic Peptide (BNP) and amino-terminal fragment of proBNP (NT-proBNP) in outpatients managed in the heart failure (HF) clinic initiated on the Angiotensin Receptor Neprilysin Inhibitor (Entresto) and directly compare the prognostic values of BNP and NT-proBNP in patients admitted with acute decompensated HF.

DETAILED DESCRIPTION:
Both natriuretic peptides (NP), namely B-type NP (BNP) and amino-terminal fragment of proBNP (NT-proBNP), have an established role in the management of patients with heart failure (HF).[1] However, the clinical utility of BNP has recently been questioned with the PARADIGM-HF trial, which demonstrated increased BNP and reduced NT-proBNP levels following the administration of Entresto, a newly approved angiotensin receptor neprilysin inhibitor (ARNI).[2.3] The increase in BNP was thought to be reflective of reduced metabolism of BNP as a result of neprilysin inhibition.[2] However, this claim was based on observations of three points in time and with wide confidence intervals.[3] In addition, there has been no attempt to demonstrate dose relationships. Furthermore, although both BNP and NT-proBNP have each been shown to predict HF readmission in hospitalized patients [1,4,5] the relative utility between the two NPs for this prediction remains unclear. We therefore hypothesize that once beyond the initiation of ARNI therapy, BNP and NT-proBNP will be equally predictive of clinical events in patients with HF.

The studies comprise of two separate protocols:

A. Outpatient Protocol - the effect of Entresto measuring the changes in the NT-proBNP and BNP test results. This protocol will be conducted on ambulatory outpatients initiating on Entresto. Patients will have blood sampling for the measurements of BNP and NT-proBNP at baseline, at the first and second up titration in dose of Entresto, and at 6 months and 1st year after starting Entresto.

B. Inpatient Protocol-predicting outcomes. This will be conducted on patients admitted for acute decompensated HF. Blood sampling for BNP and NT-proBNP will be collected in different time points (admission, hospital discharge, 30th day, 90th day, and 180th day) and measure its changes.

ELIGIBILITY:
Inclusion Criteria:

Out Patient Protocol - Patients with chronic heart failure being followed in the heart failure clinic eligible to switch angiotensin converting enzyme inhibitors (ACEI) or angiotensin receptor blockers (ARB) to ARNI (Entresto).

In Patient Protocol - Patients admitted due to acute decompensated heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-05 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Out Patient Protocol | Baseline, 2 weeks, 4 weeks, 6 months, and 12 months
  Measuring the changes with NT-prooBNP and BNP.
In Patient Protocol | Admission, discharge, 30th day post-discharge, 60th day post-discharge, and 180 days post discharge
  Measuring the changes with NT-prooBNP and BNP.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon W Moe, MD, MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moe GW, Ezekowitz JA, O'Meara E, Lepage S, Howlett JG, Fremes S, Al-Hesayen A, Heckman GA, Abrams H, Ducharme A, Estrella-Holder E, Grzeslo A, Harkness K, Koshman SL, McDonald M, McKelvie R, Rajda M, Rao V, Swiggum E, Virani S, Zieroth S, Arnold JM, Ashton T, D'Astous M, Chan M, De S, Dorian P, Giannetti N, Haddad H, Isaac DL, Kouz S, Leblanc MH, Liu P, Ross HJ, Sussex B, White M; Canadian Cardiovascular Society. The 2014 Canadian Cardiovascular Society Heart Failure Management Guidelines Focus Update: anemia, biomarkers, and recent therapeutic trial implications. Can J Cardiol. 2015 Jan;31(1):3-16. doi: 10.1016/j.cjca.2014.10.022. Epub 2014 Dec 19. PMID 25532421
- [Background] McMurray JJ, Packer M, Solomon SD. Neprilysin inhibition for heart failure. N Engl J Med. 2014 Dec 11;371(24):2336-7. doi: 10.1056/NEJMc1412654. No abstract available. PMID 25494275
- [Background] Packer M, McMurray JJ, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile M, Andersen K, Arango JL, Arnold JM, Belohlavek J, Bohm M, Boytsov S, Burgess LJ, Cabrera W, Calvo C, Chen CH, Dukat A, Duarte YC, Erglis A, Fu M, Gomez E, Gonzalez-Medina A, Hagege AA, Huang J, Katova T, Kiatchoosakun S, Kim KS, Kozan O, Llamas EB, Martinez F, Merkely B, Mendoza I, Mosterd A, Negrusz-Kawecka M, Peuhkurinen K, Ramires FJ, Refsgaard J, Rosenthal A, Senni M, Sibulo AS Jr, Silva-Cardoso J, Squire IB, Starling RC, Teerlink JR, Vanhaecke J, Vinereanu D, Wong RC; PARADIGM-HF Investigators and Coordinators. Angiotensin receptor neprilysin inhibition compared with enalapril on the risk of clinical progression in surviving patients with heart failure. Circulation. 2015 Jan 6;131(1):54-61. doi: 10.1161/CIRCULATIONAHA.114.013748. Epub 2014 Nov 17. PMID 25403646
- [Background] Logeart D, Thabut G, Jourdain P, Chavelas C, Beyne P, Beauvais F, Bouvier E, Solal AC. Predischarge B-type natriuretic peptide assay for identifying patients at high risk of re-admission after decompensated heart failure. J Am Coll Cardiol. 2004 Feb 18;43(4):635-41. doi: 10.1016/j.jacc.2003.09.044. PMID 14975475
- [Background] Maisel A, Mueller C, Adams K Jr, Anker SD, Aspromonte N, Cleland JG, Cohen-Solal A, Dahlstrom U, DeMaria A, Di Somma S, Filippatos GS, Fonarow GC, Jourdain P, Komajda M, Liu PP, McDonagh T, McDonald K, Mebazaa A, Nieminen MS, Peacock WF, Tubaro M, Valle R, Vanderhyden M, Yancy CW, Zannad F, Braunwald E. State of the art: using natriuretic peptide levels in clinical practice. Eur J Heart Fail. 2008 Sep;10(9):824-39. doi: 10.1016/j.ejheart.2008.07.014. Epub 2008 Aug 29. PMID 18760965